CLINICAL TRIAL: NCT03000998
Title: Web App Technology for Boys and Parents: Improving HPV Vaccine Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: University of New Mexico (Other); Indiana University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0310; 1R01CA210125-01A1 (NIH)
Record Dates: First submitted 2016-11-21; First posted 2016-12-22 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Human Papillomavirus Virus; HPV
Keywords: HPV; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web App Intervention Group (Experimental): The BoyVac mobile web app will be evaluated in a pair-matched group-randomized pretest-posttest controlled design. In Year 2, 30 clinics in New Mexico will be pair-matched and one member of each pair will be randomized to the intervention (mobile web app) or a usual and customary (UC) HPV vaccine adoption procedures comparison group. Clinics will be paired based on similarities in patient demographic (ethnicity and % Medicaid patients) and location (urban and rural).
  Interventions: Behavioral: Web App Intervention Group
- Usual Customary Care Group (Active Comparator): Currently in pediatric clinics in New Mexico, the HPV vaccines are offered to parents and adolescents as part of annual well-child checkups. Typically for boys aged 11-13, parents initiate this checkup as part of a back-to-school activity. As part of the well-child checkup, clinic staff (physician, physician assistant and/or nurse) talk with parents and adolescents about the recommendation that their sons or daughters receive the HPV vaccination. Well-child pediatric visits to promote good health and development are recommended for all children from infancy through adolescence by the American Academy of Pediatrics.
  Interventions: Behavioral: Usual Customary Care Group

INTERVENTIONS:
Behavioral: Web App Intervention Group — All baseline and follow-up data collection will be conducted via online surveys and a customized web portal and include parent self-reports and clinic records of vaccination of boys
  Arms: Web App Intervention Group
Behavioral: Usual Customary Care Group — Participants randomized to the usual and customary care (UC) group will receive a website with a pamphlet on HPV vaccination from the Centers for Disease Control and Prevention (CDC) in Portable Document Format (PDF) format.
  Other Names: UC
  Arms: Usual Customary Care Group

SUMMARY:
The uptake of vaccines for Human Papillomavirus (HPV) in the U.S. is far below recommended levels, particularly for adolescent boys and especially among minority families. Proposed here is a mobile web application ("mobile web app") for personal computers, smart phones, and tablet computers that will accurately inform parents and adolescent boys about the HPV vaccination and address unique concerns about its safety and effectiveness for boys. The BoyVac mobile web app will be evaluated for its ability to improve vaccine outcomes in a randomized efficacy trial with parents and adolescent boys aged 11-13 years.

DETAILED DESCRIPTION:
The President's Cancer Advisory Board and the Centers for Disease Control have called for renewed efforts in promoting vaccination for Human Papillomavirus (HPV), including vaccination for adolescent boys, because the uptake of this new vaccine remains alarmingly low. Currently, less than 15% of adolescent boys have received the HPV vaccine; thus, most of this population remains at risk for oropharyngeal, anal, and penile cancers. Many parents remain unconvinced of the safety and effectiveness of HPV vaccines, so effective and accessible messaging to improve decision-making on this vaccine is needed. Parents of adolescent boys also have different concerns about HPV vaccination than for adolescent girls, creating a need for unique health communication interventions to promote vaccine uptake among boys. Interventions also need to address the unique challenges of minority populations and populations for whom English is not the first language. A novel digital intervention will be produced and evaluated for its ability to improve HPV vaccine outcomes. Specifically, a mobile responsive web application ("mobile web app") will be created that performs similar to a mobile app but runs on a variety of computing platforms from personal desktop and laptop computers to the latest smart phones and tablet computers. Mobile web app content will be targeted to parents and adolescent boys aged 11-13 years. The specific aims are to: 1) carefully and systematically develop a mobile web app (BoyVac) for smart phones, tablet computers, and personal computers that will utilize Diffusion of Innovations principles to provide targeted information concerning HPV vaccine adoption to adolescent males and their parents, particularly minority adolescents and parents; 2) implement a comprehensive and rigorous test of the impact of the BoyVac mobile web app intervention on HPV vaccine adoption outcomes via a randomized efficacy trial (BoyVac v. usual and customary care); and 3) examine the dose-response relationships between mobile web app usage and vaccine outcomes within a components analysis. A group-randomized pretest-posttest controlled design will be implemented, recruiting 1800 pairs of parents and adolescent boys from 30 pediatric clinics (n=60 parents and boys per clinic). Parents will be surveyed at baseline, a 3-month follow-up, and a 9-month follow-up and records HPV vaccination adoption for the boys will be obtained from the clinics' medical records at the 9-month follow-up. Analyses will test the hypotheses that 1) more 11-13 year old boys in the intervention group (BoyVac mobile web app) will adopt the HPV vaccine than boys in the usual and customary care comparison group and 2) adoption of HPV vaccine will be mediated by improvements in theoretical mediators among parents in the intervention compared to the usual and customary care comparison group.

ELIGIBILITY:
Inclusion Criteria:

Adolescent boys:

1. being male
2. being 11-13 years old
3. being a patient at a participating University of New Mexico (UNM) Hospital's Envision pediatric practice
4. parental consent for testing, and
5. child assent for testing

Parents/Guardians:

1. being a parent/guardian of an eligible and participating 11-13 year old boy
2. demonstrated ability to comprehend study requirements, and
3. providing informed consent for oneself and assent for their youth's participation

Exclusion Criteria:

Adolescent boys:

1. another immediate family member is participating in the project (i.e., a sibling)
2. the participant has already received any or all doses for the HPV vaccine, or
3. the participant refuses to assent.

Parents/Guardians:

1. under the age of 18, or
2. another immediate family member is participating in the project (i.e., another parent).

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Vaccine Initiation | 1 Month
  Vaccine initiation - whether or not each boy received the HPV vaccine and the date of administration. Number of participants who received at least 1 dose.
Vaccine Adherence | 2 Months
  Vaccine Adherence - whether participants adhered to the three-dose course of the HPV vaccination or not. 2nd dose and date received. Number of participants who received at least 2 doses.
Vaccine Adherence | 4 months
  Vaccine Adherence - whether participants adhered to the three-dose course of the HPV vaccination or not. 3rd dose and date received. Number of participants who received the 3 doses.

SECONDARY OUTCOMES:
Attitudes towards vaccination in general | Baseline, 3-month follow-up, and 9-month follow-up
  Quantitative research in the form of an online survey will be conducted to examine attitudes towards vaccinations in general
Attitudes towards the HPV vaccine | Baseline, 3-month follow-up, and 9-month follow-up
  Quantitative research in the form of an online survey will be conducted to examine attitudes towards the HPV vaccine
Perception of risk due to HPV and not being vaccinated | Baseline, 3-month follow-up, and 9-month follow-up
  Quantitative research in the form of an online survey will be conducted to examine the perception of risk due to HPV and not being vaccinated.
Perception of negative and positive consequences associated with HPV vaccination | Baseline, 3-month follow-up, and 9-month follow-up
  Quantitative research in the form of an online survey will be conducted to examine the perception of negative and positive consequences associated with HPV vaccination.
Self-efficacy to make informed decisions about HPV vaccination | Baseline, 3-month follow-up, and 9-month follow-up
  Quantitative research in the form of an online survey will be conducted to examine the self-efficacy to make informed decisions about HPV vaccination
HPV knowledge | Baseline, 3-month follow-up, and 9-month follow-up
  Quantitative research in the form of an online survey will be conducted to examine the participant's knowledge about HPV
Spousal support and social normative and cultural perceptions of receiving the HPV vaccination | Baseline, 3-month follow-up, and 9-month follow-up
  Quantitative research in the form of an online survey will be conducted to examine the spousal support and social normative and cultural perceptions of receiving the HPV vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Gill Woodall, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (3):
- United States (3):
  - Klein Buendel, Inc., Golden, Colorado
  - Indiana University, Indianapolis, Indiana
  - University of New Mexico, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No